CLINICAL TRIAL: NCT03487926
Title: Naturalistic Monitoring of Microglial Activation in Inflammatory Bowel Disease
Brief Title: Microglial Activation in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Other Study IDs: 102-2016
Record Dates: First submitted 2018-01-18; First posted 2018-04-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Episode; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — N-(2-((N-(4-phenoxypyridin-3-yl)acetamido)methyl)phenoxy)ethyl fluoride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma and serum samples will be kept for analysis of genotype, peripheral inflammatory markers and protein binding.
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (3):
- Group 1 (IBD primary diagnosis): Participants have active IBD
  Interventions: Radiation: [18F]FEPPA
- Group 2( IBD + comorbid MDE): 1 [18F]FEPPA PET scan in those with IBD symptoms in the past 2 years as well present with MDE
  Interventions: Radiation: [18F]FEPPA
- Group 3-Controls: Matched for Level of Depressive Symptoms and Otherwise Healthy
  -Subjects in an otherwise healthy state with major depressive episodes, obsessive compulsive disorder, or generalized anxiety disorder will provide psychiatric diagnosis matched controls to those with IBD. Data for group three will be largely obtained from previous recent studies (it is anticipated that 95% of this data is already available).
  Interventions: Radiation: [18F]FEPPA

INTERVENTIONS:
Radiation: [18F]FEPPA — up to 3 PET Scans ([18F]FEPPA PET scans done 3 to 6 months apart, and one [11C]SL2511.88 PET scan) and 1 MRI

SUMMARY:
The purpose of this study is to monitor microglial activation in participants with inflammatory bowel disease (IBD) and investigate the relationship that exists between these patients and their risk of acquiring major depressive episodes (MDE). Patients with both IBD and MDE will be subsequently approached to participate in the study.

DETAILED DESCRIPTION:
Detailed Description:

Participants may undergo up to 3 PET Scans : [18F]FEPPA PET (for TSPO) before and 3 to 6 months later and [11C]SL25.1188 PET (for MAO-B) as well as 1 MRI scan.

The primary hypothesis is that :

1. The neuroinflammation (TSPO VT) will be increased in PFC, ACC, and insula regions in those with inflammatory bowel disease (IBD) patients compared to healthy people.
2. The neuroinflammation (TSPO VT) in PFC, ACC, and insula regions will be reduced after treatment for IBD.

The Secondary Hypothesis:

1. Elevations in neuroinflammation (TSPO VT) will be similar in those with ulcerative colitis and Crohn's disease.
2. Neuroinflammation (TSPO VT) will be greater in IBD with depression than in depression without IBD.
3. Biologics (TNFalpha antibody treatments), and fecal transplantation will be associated with greater reduction in neuroinflammation in brain than Sulfasalazine/5-Aminosalicylates.
4. MAO-B VT will be elevated in in the PFC, ACC, and insula in IBD compared to healthy controls.

There will be no alterations to standard care of patients due to participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* aside from IBD groups and common comorbidities of IBD, otherwise good physical health with no current active medical conditions.
* a lifetime diagnosis of IBD verified by medical record, which can include prescription for IBD treatment

Exclusion Criteria:

* no history of neurological illness, excluding migraine
* no use of glucocorticoid antagonists or lithium or medications that bind with affinity higher than 500nM to peripheral benzodiazepine receptors (or TSPO) in the previous two months
* no use of herbal remedies in the previous month that would be expected to influence neuroinflammation
* non-cigarette smoking
* no history of abuse of substances that affect mood and negative urine drug screens for substances of abuse including cotinine (urine drug screen is done at screening and on each PET scan day)
* no history of psychotic symptoms
* not pregnant based on a negative pregnancy test (for women)
* not breastfeeding (for women)
* no recent treatment with electroconvulsive therapy or magnetic seizure therapy in the previous 6 months
* no coagulation disorders, or anticoagulant medication use
* no presence of metal objects or implanted electrical devices in the body that would preclude MRI scanning
* no claustrophobia
* no self-reported history of fainting from blood withdrawals
* size and weight does not exceed capacity of scanner, for which size may vary and weight is 350 lbs
* no history of undergoing a number of PET scans that, including the number of PET scans under this protocol, will bring the total to more than 8 PET scans/lifetime, exceeding permissible limit for subjects participating in research set by our centre's guidelines

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community and tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
TSPO VT in prefrontal cortex, anterior cingulate cortex, and insula | within 3 to 4 weeks after initiation of screening
  Between group comparison for 3 regions in IBD compared to controls (analysis done concurrently for group effect across 3 regions)
change in TSPO VT in prefrontal cortex, anterior cingulate cortex, and insula before and after 3 to 6 months | 3 to 6 months
  Change in TSPO VT for three regions (same units for each region)
MAO-B VT in prefrontal cortex, anterior cingulate cortex, insula in IBD compared to controls | within 3 to 4 weeks after initiation of screening
  Between group comparison for 3 regions in IBD compared to controls

SECONDARY OUTCOMES:
TSPO VT in prefrontal cortex, anterior cingulate cortex, insula compared between Crohns disease and ulcerative colitis | within 3 to 4 weeks of initiating screening of subjects
  comparison of TSPO VT in 3 regions between two types of inflammatory bowel disease
TSPO VT in prefrontal cortex, anterior cingulate cortex, insula compared between IBD with MDE compared to MDE controls | within 3 to 4 weeks after initiation of screening
  Between group comparison for 3 regions in IBD compared to controls
change in TSPO VT in prefrontal cortex, anterior cingulate cortex, insula compared between naturalistic treatment with sulfasalazine/5-aminosalicylates versus other interventions like biologics or fecal transplantation | 3 to 6 months
  differential change in TSPO VT across 3 regions before and after 6 months in those receiving naturalistic treatment with sulfasalazine/5-aminosalicylates versus other naturalistic treatments of fecal transplantation or biologics

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, M.D.,PhD, Principal Investigator — Research Imaging Centre, Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Setiawan E, Wilson AA, Mizrahi R, Rusjan PM, Miler L, Rajkowska G, Suridjan I, Kennedy JL, Rekkas PV, Houle S, Meyer JH. Role of translocator protein density, a marker of neuroinflammation, in the brain during major depressive episodes. JAMA Psychiatry. 2015 Mar;72(3):268-75. doi: 10.1001/jamapsychiatry.2014.2427. PMID 25629589
- [Background] Attwells S, Setiawan E, Wilson AA, Rusjan PM, Mizrahi R, Miler L, Xu C, Richter MA, Kahn A, Kish SJ, Houle S, Ravindran L, Meyer JH. Inflammation in the Neurocircuitry of Obsessive-Compulsive Disorder. JAMA Psychiatry. 2017 Aug 1;74(8):833-840. doi: 10.1001/jamapsychiatry.2017.1567. PMID 28636705
- [Background] Holmes SE, Hinz R, Conen S, Gregory CJ, Matthews JC, Anton-Rodriguez JM, Gerhard A, Talbot PS. Elevated Translocator Protein in Anterior Cingulate in Major Depression and a Role for Inflammation in Suicidal Thinking: A Positron Emission Tomography Study. Biol Psychiatry. 2018 Jan 1;83(1):61-69. doi: 10.1016/j.biopsych.2017.08.005. Epub 2017 Aug 12. PMID 28939116
- [Background] Li H, Sagar AP, Keri S. Translocator protein (18kDa TSPO) binding, a marker of microglia, is reduced in major depression during cognitive-behavioral therapy. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Apr 20;83:1-7. doi: 10.1016/j.pnpbp.2017.12.011. Epub 2017 Dec 19. PMID 29269262